CLINICAL TRIAL: NCT07122687
Title: A Phase II Study Evaluating the Efficacy and Safety of IBI363 Combined With Chemotherapy or Pembrolizumab Combined With Chemotherapy as Neoadjuvant Therapy in Resectable Stage IB-III Non-Squamous Non-Small Cell Lung Cancer
Brief Title: IBI363 Combined With Chemotherapy or Pembrolizumab Combined With Chemotherapy as Neoadjuvant Therapy in Resectable Stage IB-III Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363C201
Record Dates: First submitted 2025-06-24; First posted 2025-08-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Resectable Stage IB-III Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Cisplatin; Carboplatin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI363 (Experimental): Neoadjuvant Treatment period: up to 3 cycles of IBI363 plus platinum-based chemotherapy prior to surgery.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: IBI363; Drug: Carboplatin
- Keytruda (Active Comparator): Neoadjuvant Treatment period: up to 3 cycles of Keytruda plus platinum-based chemotherapy prior to surgery.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Keytruda

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 D1 IV Q3W
Drug: Cisplatin — 75 mg/m2 D1 IV Q3W
Drug: IBI363 — 1.5 mg/kg D1 IV Q3W
  Arms: IBI363
Drug: Carboplatin — AUC 5 mg/ml/min D1 IV Q3W
Drug: Keytruda — 200mg D1 IV Q3W
  Arms: Keytruda

SUMMARY:
This study is a randomized, open-label Phase 2 study to compare the efficacy and safety of IBI363 Combined with Chemotherapy or Pembrolizumab Combined with Chemotherapy as Neoadjuvant Therapy in Resectable Stage IB-III Non-Squamous Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females, age ≥18 years and ≤75 years;
2. Histologically or cytologically confirmed primary non-squamous NSCLC:

   * Stage IB, II, IIIA or IIIB (N2) NSCLC (per AJCC8);
   * No administration of any anti-NSCLC therapy in the pre-operative period;
   * Be able to undergo the radical resection; Pulmonary function capacity capable of tolerating the proposed lung resection according to the surgeon.
3. Participants without EGFR mutations or ALK translocation;
4. At least 1 measurable lesion per RECISIT v1.1;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1;
6. Adequate organ function confirmed at screening period.

Exclusion Criteria:

1. Histologically confirmed the presence of small cell lung cancer, neuroendocrine carcinoma, sarcoma, salivary gland tumor, and mesenchymal tumor components, or mixed NSCLC with predominant squamous cell carcinoma features;
2. Tumor invasion of surrounding important structures, which is symptomatic or medical intervention indicated;
3. Pancoast tumor;
4. Malignant tumor nodule in the contralateral lung lobe;
5. Participants with known or suspected brain metastases or other distant metastases;
6. Participants who received Chinese herbal medicines, proprietary Chinese medicines with anti-tumor indications, or immunomodulatory drugs within 2 weeks prior to the first dose of the study drug;
7. Participants with a condition requiring systemic treatment with corticosteroids or is receiving any other form of immunosuppressive therapy within 7 days prior the first dose of the study drug;
8. History of any arterial thromboembolic event within 6 months prior to the first dose of the study drug;
9. History of deep vein thrombosis, pulmonary embolism, or any other serious venous thromboembolism within 3 months prior to the first dose of study drug;
10. History of pneumonitis requiring corticosteroid therapy, or history of clinically significant lung diseases or who are suspected to have these diseases by imaging during the screening period;
11. Active or uncontrolled diseases or conditions;
12. History of immunodeficiency disease;
13. Participants with active autoimmune disease requiring systemic treatment within 2 years prior to the first dose of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  pCR rate is defined as no residual invasive viable tumor in both the primary tumor (lung) and the sampled lymph nodes after neoadjuvant therapy.
Safety parameters: the incidence of all adverse events (AEs) | up to 90 days after the last dose
Safety parameters: the incidence of treatment-emergent adverse events (TEAEs) | up to 90 days after the last dose
Safety parameters: the incidence of immune-related adverse events (irAEs) | up to 90 days after the last dose
Safety parameters: the incidence of adverse events of special interest (AESIs) | up to 90 days after the last dose
Safety parameters: the incidence of serious adverse events (SAE) | up to 90 days after the last dose
Safety parameters: the relatedness of infusion-related reactions (IRRs) to the investigational product and their severity | up to 90 days after the last dose
Safety parameters: the surgery delay rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
Proportion of subjects with abnormal and clinically significant results including routine blood tests, blood biochemical tests, coagulation tests,, routine urine tests, pregnancy tests，ECG, etc | up to 90 days after the last dose

SECONDARY OUTCOMES:
Event Free Survival (EFS) | Up to approximately 5 years
  EFS is defined as the time from the first dose to the first determination by the investigator with RECIST v1.1 of inoperable disease progression, postoperative local recurrence or distant metastasis, development of another primary tumor, or death from any cause, whichever occurred first.
Major Pathological Response (mPR) Rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  mPR rate is defined as ≤ 10% residual invasive viable tumor in both the primary tumor (lung) and the sampled lymph nodes after neoadjuvant therapy.
Objective Response Rate （ORR）Rate | Up to approximately 5 years
  ORR is defined as the proportion of subjects assessed by the investigators as achieving complete response (CR) or partial response (PR) according to the RECIST v1.1 criteria.
Disease Control Rate (DCR) Rate | Up to approximately 5 years
  ORR is defined as the proportion of subjects assessed by the investigators as achieving complete response (CR) 、partial response (PR) or stable Disease（SD） according to the RECIST v1.1 criteria.
R0 resection rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  R0 resection rate is defined as negative margins, systematic lymph node dissection or sampling, and tumor-negative highest mediastinal lymph nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Cancer Hospital and Institute, Shenyang, Liaoning, China